CLINICAL TRIAL: NCT00634504
Title: An Open-Label Study to Assess the Pharmacokinetics of Leucovorin in Patients Receiving High Dose Methotrexate, With or Without Voraxaze Treatment
Brief Title: Open-label Leucovorin Pharmacokinetic Study in Patients Receiving High Dose Methotrexate With or Without Voraxaze
Acronym: LVPK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR001-CLN-pro017
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Osteosarcoma; Leukemia; Lymphoma
Keywords: high dose methotrexate; Voraxaze; leucovorin; delayed elimination; methotrexate toxicity; rescue; renal insufficiency
MeSH Terms: conditions — Osteosarcoma; Leukemia; Lymphoma; Renal Insufficiency | interventions — glucarpidase; Methotrexate; Leucovorin; gamma-Glutamyl Hydrolase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): High-dose methotrexate, leucovorin, and Voraxaze
  Interventions: Drug: glucarpidase, high-dose methotrexate, leucovorin
- B (Active Comparator): High-dose methotrexate and leucovorin without Voraxaze (glucarpidase)
  Interventions: Drug: high-dose methotrexate, leucovorin

INTERVENTIONS:
Drug: glucarpidase, high-dose methotrexate, leucovorin — single intravenous dose
  Other Names: Voraxaze, carboxypeptidase G2, high dose methotrexate, leucovorin
  Arms: A
Drug: high-dose methotrexate, leucovorin — standard of care, leucovorin every 6 hours
  Other Names: HDMTX, LV
  Arms: B

SUMMARY:
The purpose of this study is to investigate whether the administration of Voraxaze reduces exposure to leucovorin and its active metabolite to below the level achieved in patients who have not received Voraxaze.

ELIGIBILITY:
Inclusion Criteria:

* Receiving High-dose methotrexate (HDMTX) with or without risk of methotrexate (MTX) toxicity, impaired renal function, and delayed MTX elimination
* Require intravenous leucovorin

Exclusion Criteria:

* Arm A only: allergic reactions to lactose
* Arm A only: hereditary fructose or galactose intolerance
* Arm B only: delayed elimination of MTX

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Saunders, MD, Study Chair; Suzanne Kincaid, CCRA, Study Director — BTG International Inc.
Locations (25):
- United States (25):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Good Samaritan Hospital, Los Angeles, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Los Angeles, California
  - Oakland's Children's Hospital, Oakland, California
  - Stanford University Medical Center & Lucile Packard Children's Hospital, Palo Alto, California
  - California Pacific Medical Center, San Francisco, California
  - Children's Hospital for Cancer & Blood Disorders, Aurora, Colorado
  - St. Joseph's Hospital, Tampa, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University of Massachusetts - Umass Memorial Medical Center, Worcester, Massachusetts
  - University of MS Medical Center, Jackson, Mississippi
  - University of Missouri-Columbia, Columbia, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - ECU Brody School of Medicine, Greenville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Huntsman Cancer Center, Salt Lake City, Utah
  - Children's Hospital and Regional Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- A (High-dose Methotrexate, Leucovorin, and Glucarpidase): Drug: High-dose methotrexate (HDMTX) and leucovorin (LV) with a single bolus intravenous injection of 50 units/kg glucarpidase over 5 minutes.
  HDMTX followed by intravenous LV administered at doses recommended in the clinical treatment protocols.
  LV doses administered as recommended in the package insert for Leucovorin Calcium USP for patients with delayed early MTX elimination and/or evidence of acute renal injury, and should be based upon the pre-glucarpidase MTX concentration. LV doses are maintained for at least 48 hours after dosing with glucarpidase. After this it may be administered at doses recommended in the clinical treatment protocols and existing labeling for LV based on post-Voraxaze MTX concentrations. Patients required IV LV rescue therapy with either ≥15 mg or ≥10 mg/m2 every 6 hours.
  Other Names:
  Voraxaze, carboxypeptidase G2, high dose methotrexate, leucovorin
- B (High-dose Methotrexate and Leucovorin Without Glucarpidase): High-dose methotrexate (HDMTX) and leucovorin (LV) without glucarpidase
  HDMTX followed by intravenous LV should be administered at doses recommended in the clinical treatment protocols and as per standard of care. LV should be given every 6 hours at a dose of ≤25 mg/m2.
Period: Overall Study
Arm/Group | A (High-dose Methotrexate, Leucovorin, and Glucarpidase) | B (High-dose Methotrexate and Leucovorin Without Glucarpidase)
Started | 11 | 9
Completed | 10 | 9
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- A (High-dose Methotrexate, Leucovorin, and Glucarpidase): High-dose methotrexate, leucovorin, and glucarpidase
  glucarpidase, high-dose methotrexate, leucovorin: single intravenous dose
- B (High-dose Methotrexate and Leucovorin Without Glucarpidase): High-dose methotrexate and leucovorin without glucarpidase
  high-dose methotrexate, leucovorin: standard of care, leucovorin every 6 hours
- Total: Total of all reporting groups
Arm/Group | A (High-dose Methotrexate, Leucovorin, and Glucarpidase) | B (High-dose Methotrexate and Leucovorin Without Glucarpidase) | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (22.07) | 12.6 (7.84) | 20.2 (18.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 7 | 13
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Pre-glucarpidase (Arm A) or Pre-LV (Arm B) methotrexate plasma conc (umol/L) [Mean (Standard Deviation); unit: micromol/L] | 34.58 (48.59) | 6.49 (11.00) | 21.94 (21.94)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Leucovorin
Description: Geometric mean (6S)-leucovorin area under the plasma concentration vs. time curve from time 0 to the 3-hour time point.
Time Frame: 5 minutes, 30 minutes, 1 hour, 2 hours and 3 hours post-LV administration
Population: 3 participants were excluded from the PK population (all from Arm A), hence why the total participants is 17, not 20.
Measure: Geometric Mean (95% Confidence Interval); unit: micromol x hour/L
Arm/Group | A (High-dose Methotrexate, Leucovorin, and Glucarpidase) | B (High-dose Methotrexate and Leucovorin Without Glucarpidase)
Number analyzed (Participants) | 8 | 9
micromol x hour/L | 6.43 [2.89 to 14.32] | 1.13 [0.72 to 1.75]

ADVERSE EVENTS:
Arm/Group | A (High-dose Methotrexate, Leucovorin, and Glucarpidase) | B (High-dose Methotrexate and Leucovorin Without Glucarpidase)
Serious Adverse Events (participants affected / at risk) | 3/11 | 0/9
Other Adverse Events (participants affected / at risk) | 7/11 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (High-dose Methotrexate, Leucovorin, and Glucarpidase) (N=11) | B (High-dose Methotrexate and Leucovorin Without Glucarpidase) (N=9)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (High-dose Methotrexate, Leucovorin, and Glucarpidase) (N=11) | B (High-dose Methotrexate and Leucovorin Without Glucarpidase) (N=9)
neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 3 (3) | 0 (0)
flushing (Vascular disorders) | 1 (1) | 0 (0)
hemoglobin decreased (Investigations) | 2 (2) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
serum creatinine increased (Investigations) | 1 (1) | 0 (0)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypomagnesmia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
mucosal inflammation (General disorders) | 2 (2) | 0 (0)
pyrexia (General disorders) | 1 (1) | 0 (0)
burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
hypoesthesia (Nervous system disorders) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0)
paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No